CLINICAL TRIAL: NCT06628050
Title: Post-market Observational Study of the ORIGIN® PS Modular Total Knee Prosthesis and Associated Instruments
Brief Title: ORIGIN® PS Modular & Associated Instruments
Status: Active, not recruiting | Type: Observational
Sponsor: Symbios Orthopedie SA (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN-G-013
Record Dates: First submitted 2024-05-07; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Total Knee Replacement
Keywords: TKA; ORIGIN; Prosthesis; Postero-stabilized; Modular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ORIGIN® PS Modular devices — Consecutive eligible subjects have been included which have been treated with the ORIGIN® PS Modular devices.

SUMMARY:
The study objective is to evaluate safety and performance of the ORIGIN® PS (postero-stabilized) Modular devices and associated instruments, more precisely to evaluate safety by the proportion of patients requiring a revision (i.e. revision rate) at 2-6 months, 1y and 2y post-procedure and to evaluate performance by means of a Knee Society Score (KSS) Score at 2-6 months, 1y and 2y post procedure.

The hypothesis raised for this study, regarding the scoring, is that patients will experience a marked improvement in the natural feel of the prosthesis during the first year after the surgery, and slightly significant improvement at the following interval of 2 years. The overall patient satisfaction is expected to be improved after 2 years follow-up with ORIGIN® PS Modular.

DETAILED DESCRIPTION:
The study is ambispective, post market, non-comparative, non-randomized, multicentric and observational in which 200 patients will be enrolled to evaluate the safety and performance of the ORIGIN® PS Modular devices and associated instruments.

Patients will be included in the study during 18 months (inclusion window) and followed-up for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 years of age.
* Patient, or if applicable, his or her guardian or legal representative, willing to give informed consent.
* Clinically indicated for first intention total knee replacement.
* Geographically stable and willing to return for all follow-up visits or, at a minimum, to complete the patient self-report score.

Exclusion Criteria:

* Vulnerable subject (as defined in ISO-14155)
* Acute or chronic, local or systemic infection,
* Muscular, ligamental, neurological, psychological or vascular deficits,
* Bone destruction or poor bone quality likely to affect implant stability.
* Any concomitant condition likely to affect implant integration or function,
* Allergy or hypersensitivity to any of the materials used,
* For devices in CoCr Mo (ISO 5832/4): renal and hepatic impairment,
* Hip Knee Ankle (HKA) angle < 165° or > 195°,
* Severe collateral ligament deficiency (requiring a more constrained prosthesis),
* Major anatomical deformities,
* Severe flexion contracture or severe recurvatum,
* Revision of a partial or total knee prosthesis,
* Non-extractible material (e.g., screw, plate, intramedullary nail, osteosynthesis material) which can create a conflict with any component of the prosthesis,
* Distal and/or posterior and/or anterior femoral bone loss which exceeds the femoral component thickness,
* Proximal tibial bone loss which exceeds the tibial component thickness (tibial tray + tibial insert),
* Bone degradation requiring an anchoring stem for femoral component

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have provided consent for the collection of their data and met the protocol eligibility criteria will be enrolled into this observational non-comparative ambispective multicentric study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-04-18 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Evaluate safety by the proportion of required revisions | 2 years post-op procedure
  Proportion of patients requiring a revision at each follow-up visit (surgery, 2-6 months, 1- and 2 years). The revision rate is consistent with the state of the art - Orthopaedic Data Evaluation Panel (ODEP) benchmark system (revision rate not higher than 2.5% to 3.5% at 1 year, 4% to 6% at 5 years and 5% to 7% at 10 years).
Evaluate performance | 2 years post-op procedure
  Evaluate performance by means of a Knee Society Score (KSS) and a KSS Function score.
  It aims to reach a KSS Knee score of at least 85,5 / 100 points and a KSS Function score of at least 72,5 / 100 points.

SECONDARY OUTCOMES:
Evaluate the success of the surgical procedure by means of a surgeon satisfaction questionnaire. | Perioperative
  Surgeon satisfaction: during surgery, the surgeon will assess safety and performance of the associated Instrumentation and implants. The criteria of evaluation of the satisfaction are: Very satisfied - satisfied - unsatisfied - very unsatisfied. Each surgical step is evaluated for each instrument and implant component used by the surgeon. These data will be collected in the case report form based on surgeon satisfaction questionnaire and will be used in clinical evaluation of ORIGIN® PS Modular.
Evaluate safety by analyzing the occurencies of adverse events. | Perioperative and 2 years post-op procedure
  * Evaluate the intraoperative difficulties and complications (the rate should not be higher than 1,8% according to the state of the art).
  * Evaluate post-operative complications during the entire study period.
  * Evaluate the safety of the modular tibial stem by analysing the revision rate for aseptic tibial loosening at each follow-up visit (surgery, 2-6 months, 1 year and 2 years) with a maximum revision rate for aseptic loosening of 5.3% for first intention total knee replacements as cited in the knee joint registries.
Patient Quality of Life by means of the FJS score | 2 years post-op procedure
  Assess patients' ability to forget their knee in the short term after surgery, as measured by the "Forgotten Knee Score" (FJS-12: from 0 to 100 points, meaning that "0" is worst case and "100" the best).

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Polyclinique Medipole Saint Roch, Cabestany
  - Clinique Juge, Marseille

IPD SHARING:
Plan to Share IPD: No